CLINICAL TRIAL: NCT03213015
Title: Correlation Between the Amplitude of Ankle Dorsiflexion and Occurrence of Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Filipe Abdalla dos Reis (Other)
Responsible Party: Sponsor-Investigator, Filipe Abdalla dos Reis, Principal Investigator and Clinical Professor, Universidade Anhanguera
Organization: Universidade Anhanguera (Other)
Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2.128.451
Record Dates: First submitted 2017-07-04; First posted 2017-07-11 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: confiability; ankle; patellofemoral pain syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Measurement of ankle dorsiflexion ROM (range of motion) with iHand app (smartphone)
  Interventions: Diagnostic Test: Ankle dorsiflexion measurement

INTERVENTIONS:
Diagnostic Test: Ankle dorsiflexion measurement — It was used the test with WB, called Lunge Test, in which each evaluator marked a point 15 cm distal to the anterior tuberosity of the tibia (TAT) with a felt tip pen. After that the smartphone (app iHand) will be placed at this point. Between each measurement, the mark was removed with alcohol 70% The demarcated point served as a guide for positioning the smartphone. In order to standardize the smartphone positioning, BHome (home button on the iPhone), was aligned with the TAT pen mark. To ensure the same distance from the foot to the test, the distance of the hallux to the wall was measured (tape measure), recorded and reused for each test.

SUMMARY:
The aim of this study was to verify the clinical reliability of ankle dorsiflexion range of motion (ADROM) measurement with weight bearing (WB) using an app on the smartphone (iHand) and to verify if there is correlation between the limitation of the ADROM and the PFP.

DETAILED DESCRIPTION:
The change in lower extremity movement pattern has been previously associated with severe knee disorders, including anterior cruciate ligament rupture, patellar tendinopathy, iliotibial band syndrome, and patellofemoral pain (PFP). The aim of this study was to verify the clinical reliability of ankle dorsiflexion range of motion (ADROM) measurement with weight bearing (WB) using an app on the smartphone (iHand) and to verify if there is correlation between the limitation of the ADROM and the PFP.

ELIGIBILITY:
Inclusion Criteria:

* volunteers with a history of patelofemoral pain
* presence of image (lesion) in cartilage tissue in Nuclear Magnetic Resonance
* knee dynamic valgus during the single leg squat test and step down test (clinical tests)

Exclusion Criteria:

* acute knee lesion
* acute ankle lesion
* surgical procedures before six months ago

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2017-03-25 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Ankle Dorsiflexion Degrees | 1 day
  We will evaluate the ankle range of motion (dorsiflexion) with app (iHand) in smartphone. The measurement will be in degree.

CONTACTS AND LOCATIONS:
Locations (1):
- Filipe Abdalla, Campo Grande, Mato Grosso do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dill KE, Begalle RL, Frank BS, Zinder SM, Padua DA. Altered knee and ankle kinematics during squatting in those with limited weight-bearing-lunge ankle-dorsiflexion range of motion. J Athl Train. 2014 Nov-Dec;49(6):723-32. doi: 10.4085/1062-6050-49.3.29. PMID 25144599